CLINICAL TRIAL: NCT01819337
Title: The Influence of Preoperative Cardiopulmonary Capacity Mesured in MET's (Metabolic Equivalents) on the Perioperative Lactate Level
Brief Title: The Influence of Preoperative Cardiopulmonary Capacity on the Perioperative Lactate Level
Status: Completed | Type: Observational
Sponsor: University of Witten/Herdecke (Other)
Responsible Party: Principal Investigator, Armin Zagler, MD, University of Witten/Herdecke
Other Study IDs: Lactate1
Record Dates: First submitted 2013-02-08; First posted 2013-03-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Sensitivity Training Groups; Complication, Cardio-respiratory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to identify if there exists a correlation between the preoperative cardiopulmonary capacity - measured in MET's - and the perioperative lactate serum level.

DETAILED DESCRIPTION:
The determination of the cardiopulmonary (c/p) capacity is very important for the evaluation of every patient undergoing surgery. The ability to climb at least two flight of stairs is seen to be an acceptable c/p capacity for surgery. There are several ways to evaluate the fitness of patients. A common method to estimate the cardiopulmonary capacity is defining patients through the MET's (metabolic equivalents) scale. MET's can be defined relatively easy through a simple questionnaire. Patients with a reduced c/p capacity have less than 4 MET's, patients with a relatively good c/p capacity have 4-10 MET's and patients with a excellent c/p capacity have more than 10 MET's.

The lactate level in blood serum is a common parameter to asses anaerobic metabolism in patients. A high lactate level correlates with higher mortality rates and outcome.

To yet it is not clear if there exists a correlation between the preoperative cardiopulmonary capacity measured in MET's and the perioperative lactate level. We hypothysed that patients with a reduced cardiopulmonary capacity are associated with higher perioperative lactate levels, as these group of patients compensate the stressors operation/anesthesia less than patients with a good c/p capacity.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years

Exclusion Criteria:

* Cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing elective/urgent or emergency surgery
Sampling Method: Non-Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 2013-03; Primary Completion 2013-04 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
lactate - venous blood gas analysis | venous lactate will be measured at anaesthesia induction and anesthesia termination - the average time frame is 2 hours
  mmol/l

SECONDARY OUTCOMES:
icu in hospital mortality | icu patients will be followed over their hospital stay over a maximum period of 6 months
hemoglobin - venous blood gas analysis | hemoglobin will be measured at anaesthesia induction and anesthesia termination - the average time frame is 2 hours
  g/dl
icu ventilation time | icu patients will be followed over their hospital stay over a maximum period of 6 months
  hours/days

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Schneider, Prof., Study Chair — Dept. Anaesthesiology
Locations (1):
- Helios Klinikum Wuppertal, Wuppertal, North Rhine-Westphalia, Germany